CLINICAL TRIAL: NCT04827836
Title: Pain Control and Subconjunctival Hemorrhage Size After Intravitreal Injection Using Cooled Anesthetic Eye Drops and Antiseptics: A Double-Blind Randomized Controlled Trial
Brief Title: Pain Control and Subconjunctival Hemorrhage Size After Intravitreal Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Oriel Spierer, Director of the Pediatric Ophthalmology Unit, Wolfson Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 0255-20-WOMC
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-07

CONDITIONS: Intravitreal Injection; Pain; Subconjunctival Hemorrhage
Keywords: Intravitreal injection; Pain; Subconjunctival Hemorrhage; Bevacizumab; Eye drops
MeSH Terms: conditions — Pain | interventions — Povidone-Iodine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A - Room-temperature eye drops and povidone-iodine (No Intervention): Participants will receive a standardized topical anesthesia protocol of oxybuprocaine hydrogen chloride (HCl) 0.4% and lidocaine HCl 2% eye drops. Each drop will be instilled 3 times (one drop): At 10 minutes, 5 minutes, and just before the injection. Before the injection patients will receive cul-de-sac 5% povidone-iodine (3 drops) and the peri-ocular skin will be disinfected using a 10% povidone-iodine. A standard intravitreal injection of bevacizumab, 1.25 mg/0.05 ml will be performed through the pars plana with a 30-gauge needle, 3.5 mm from the corneal limbus, at the superior-temporal quadrant. Following the injection, a cotton swab absorbed with 5% povidone-iodine will be applied to the injection site.
- Cohort B - Cooled eye drops and povidone-iodine (Experimental): Participants will receive the same treatment as cohort A, using cooled eye drops and povidone-iodine (5 degree Celsius).
  Interventions: Procedure: Cooled eye drops and povidone-iodine

INTERVENTIONS:
Procedure: Cooled eye drops and povidone-iodine — Cooled oxybuprocaine HCl 0.4% and lidocaine HCl 2% eye drops and cooled povidone-iodine (cul-de-sac 5% povidone-iodine and 10% povidone-iodine).
  Arms: Cohort B - Cooled eye drops and povidone-iodine

SUMMARY:
Intravitreal injections (IVI) are the mainstay of treatment modality in many ophthalmologic diseases including neovascular age-related macular degeneration (AMD), diabetic retinopathy and retinal vascular occlusions. Patients endure monthly IVI for several years. Although standardized topical anesthesia protocols are being carried out, many still suffer from pain during and after the procedure. Previous studies at the investigators clinic have demonstrated that alpha-agonist eye drops and cool eye compresses can be successfully used in order to reduce pain levels when administered prior to IVI. In the current research, the investigators wish to study whether cooled anesthetic eye drops and antiseptics can be utilized as well to reduce the pain and subconjunctival hemorrhage caused by bevacizumab IVI.

ELIGIBILITY:
Inclusion Criteria:

* Participants over the age of 18 years, receiving Bevacizumab IVI who are capable of signing a written informed consent form obtained under the Declaration of Helsinki.

Exclusion Criteria:

* No consent to participate in the study.
* Incapability of signing a written informed consent form.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-07-11 (Actual); Primary Completion 2021-12-27 (Actual); Study Completion 2021-12-27 (Actual)

PRIMARY OUTCOMES:
Participant's discomfort after intravitreal injection (IVI) as assessed by the visual analog scale (VAS) and pain sensitivity questionnaire (PSQ). | Minute 1
  The VAS will be used to measure participant's discomfort, itching, burning, and pain (the VAS scale ranges from 0-10, '0' being no pain at all and '10' being the most severe pain). For each participant, tolerability score will be calculated by averaging the participant's discomfort, itching, burning, and pain. To estimate the participant's baseline pain scores, a self-reported pain sensitivity questionnaire, the PSQ, will be used prior to IVI. This is a validated 17-item questionnaire designed to assess an individual's baseline pain sensitivity.
Participant's discomfort after intravitreal injection (IVI) as assessed by the visual analog scale (VAS) and pain sensitivity questionnaire (PSQ). | Minute 10
  The VAS will be used to measure participant's discomfort, itching, burning, and pain (the VAS scale ranges from 0-10, '0' being no pain at all and '10' being the most severe pain). For each participant, tolerability score will be calculated by averaging the participant's discomfort, itching, burning, and pain. To estimate the participant's baseline pain scores, a self-reported pain sensitivity questionnaire, the PSQ, will be used prior to IVI. This is a validated 17-item questionnaire designed to assess an individual's baseline pain sensitivity.
Participant's discomfort after intravitreal injection (IVI) as assessed by the visual analog scale (VAS) and pain sensitivity questionnaire (PSQ). | Hour 2
  The VAS will be used to measure participant's discomfort, itching, burning, and pain (the VAS scale ranges from 0-10, '0' being no pain at all and '10' being the most severe pain). For each participant, tolerability score will be calculated by averaging the participant's discomfort, itching, burning, and pain. To estimate the participant's baseline pain scores, a self-reported pain sensitivity questionnaire, the PSQ, will be used prior to IVI. This is a validated 17-item questionnaire designed to assess an individual's baseline pain sensitivity.
Participant's discomfort after intravitreal injection (IVI) as assessed by the visual analog scale (VAS) and pain sensitivity questionnaire (PSQ). | Hour 24
  The VAS will be used to measure participant's discomfort, itching, burning, and pain (the VAS scale ranges from 0-10, '0' being no pain at all and '10' being the most severe pain). For each participant, tolerability score will be calculated by averaging the participant's discomfort, itching, burning, and pain. To estimate the participant's baseline pain scores, a self-reported pain sensitivity questionnaire, the PSQ, will be used prior to IVI. This is a validated 17-item questionnaire designed to assess an individual's baseline pain sensitivity.

SECONDARY OUTCOMES:
Participant's subconjunctival hemorrhage (SCH) size after intravitreal injection (IVI) as evaluated by a slit lamp examination. | Minute 10
  SCH size following IVI will be photographed using a slit lamp camera at a uniform magnification and quantified using an image analysis software.

CONTACTS AND LOCATIONS:
Overall Officials: Oriel Spierer, MD, Principal Investigator — Wolfson Medical Center
Locations (1):
- Wolfson Medical Center, Holon, Central District, Israel